CLINICAL TRIAL: NCT07014202
Title: Comparing Consolidation Radiotherapy Versus No Radiotherapy for Oligoresidual Disease After First-line Chemotherapy Plus Immunotherapy in Advanced Non-Small Cell Lung Cancer: A Prospective, Randomized Controlled Phase II Clinical Trial
Brief Title: Consolidation Radiotherapy vs. Observation in Oligoresidual Advanced Non-Small Cell Lung Cancer After Chemo-Immunotherapy
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Cancer Institute and Hospital, Chinese Academy of Medical Sciences (Other)
Responsible Party: Principal Investigator, Zhijie Wang, Professor, Cancer Institute and Hospital, Chinese Academy of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCC4839
Record Dates: First submitted 2025-05-26; First posted 2025-06-10 (Actual); Last update posted 2025-07-30 (Actual); Status verified 2025-05

CONDITIONS: Non-Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Immunotherapy; Radiotherapy; Maintenance

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Maintenance therapy combined with radiotherapy group (Experimental): Radiotherapy Protocol:
  Target all residual primary lesions and all metastatic sites (pulmonary, hepatic, osseous, lymphadenopathy). Fractionation determined by treating physician after multidisciplinary consultation. For lesions near critical organs, appropriate fractionation/total doses selected per clinical situation.
  Maintenance Therapy Protocol:
  Based on latest National Comprehensive Cancer Network (NCCN)/Chinese Society of Clinical Oncology(CSCO) guidelines for stage IV non-small cell lung cancer (NSCLC). For lung adenocarcinoma: Following 4-6 cycles of first-line therapy (pemetrexed+platinum+immunotherapy) Maintenance: Pemetrexed (500mg/m²) + pembrolizumab 200mg IV q3w. Duration: Maximum 24 months (until week 96, disease progression, unacceptable toxicity, consent withdrawal, or other termination criteria). All trial patients receive immunotherapy maintenance
  Interventions: Combination Product: Immunotherapy (with or without chemotherapy) maintenance therapy combined with radiotherapy
- Maintenance therapy (Active Comparator): Based on latest NCCN/CSCO guidelines for stage IV NSCLC. For lung adenocarcinoma: Following 4-6 cycles of first-line therapy (pemetrexed+platinum+immunotherapy) Maintenance: Pemetrexed (500mg/m²) + pembrolizumab 200mg IV q3w. Duration: Maximum 24 months (until week 96, disease progression, unacceptable toxicity, consent withdrawal, or other termination criteria). All trial patients receive immunotherapy maintenance
  Interventions: Drug: Immunotherapy (with or without chemotherapy) maintenance therapy

INTERVENTIONS:
Combination Product: Immunotherapy (with or without chemotherapy) maintenance therapy combined with radiotherapy — Immunotherapy (with or without chemotherapy) maintenance therapy combined with radiotherapy in patients with advanced NSCLC who have not progressed after 4-6 cycles of first-line platinum-containing chemotherapy combined with immunotherapy and who have an oligo-residual status confirmed by PETCT.
  Arms: Maintenance therapy combined with radiotherapy group
Drug: Immunotherapy (with or without chemotherapy) maintenance therapy — Immunotherapy (with or without chemotherapy) maintenance therapy in patients with advanced NSCLC who have not progressed after 4-6 cycles of first-line platinum-containing chemotherapy combined with immunotherapy and who have an oligo-residual status confirmed by PETCT.
  Arms: Maintenance therapy

SUMMARY:
This clinical study investigates whether adding local radiation therapy (radiotherapy) to standard maintenance therapy benefits patients with advanced non-small cell lung cancer (NSCLC) who have a limited number of residual tumors after initial treatment.

The primary objective is to determine if adding targeted radiation therapy to residual lesions prolongs progression-free survival in NSCLC patients with "oligo-residual lesions" (5 or fewer tumors in no more than 3 organs) following first-line chemoimmunotherapy. Researchers hypothesize that combination therapy will slow cancer progression more effectively than maintenance therapy alone.

Eligible participants include adults (18+) with advanced NSCLC who have completed 4-6 cycles of first-line chemoimmunotherapy, show limited residual disease on Positron Emission Tomography-Computed Tomography (PET-CT), and lack specific genetic mutations (Epidermal Growth Factor Receptor [EGFR], Anaplastic Lymphoma Kinase [ALK], etc.).

Patients will be randomized into two groups:

Experimental: Continuation of maintenance therapy (immunotherapy alone or with chemotherapy) plus local radiotherapy to all residual tumors Control: Continuation of maintenance therapy only

The study aims to answer:

Primary: Does adding radiotherapy slow cancer progression more effectively? Secondary: Does it improve overall survival, control residual disease, and what are its effects on safety and quality of life?

Participants will:

Be randomly assigned to a treatment group Receive their designated treatment Undergo regular check-ups and imaging scans Complete quality of life questionnaires Potentially provide blood samples for research This research will help determine optimal treatment approaches for this specific patient population to improve outcomes and quality of life.

DETAILED DESCRIPTION:
The purpose of this clinical study is to find out whether the addition of local radiation therapy (radiotherapy) after standard chemotherapy and immunotherapy is better than continuing maintenance therapy alone for patients with specific types of advanced lung cancer .

Study Objectives and Hypotheses:

The primary objective is to see if the addition of radiation therapy to target residual lesions will prolong the time that a patient's cancer does not get worse (progression-free survival) in patients with advanced non-small cell lung cancer (NSCLC) who have a limited number of tumors (known as "oligo-residual lesions") after receiving first-line chemotherapy in combination with immunotherapy . The researchers hypothesized that patients who receive maintenance therapy plus radiation therapy will have their cancer progress more slowly than patients who receive only maintenance therapy .

Study Population:

This study is for adult patients 18 years of age and older who have been diagnosed with advanced non-small cell lung cancer . These patients have received 4 to 6 cycles of first-line chemotherapy in combination with immunotherapy and have a limited number of tumor lesions on post-treatment imaging (PET-CT) (no more than 5 residual lesions involving no more than 3 organs) and no specific genetic mutations (e.g., Epidermal Growth Factor Receptor [EGFR], Anaplastic Lymphoma Kinase [ALK], etc.).

Study Methods:

Eligible patients will be randomly assigned to one of two groups :

Experimental group: continuation of maintenance therapy (either immunotherapy or chemotherapy combined with immunotherapy, depending on the previous regimen) and local radiotherapy to all residual tumor lesions.

Control group: Continuation of maintenance therapy only.

Key questions to be answered by the study:

Primary question: is the addition of local radiotherapy more effective in slowing cancer progression than maintenance therapy alone in this group of lung cancer patients? Secondary questions include: Does the addition of radiotherapy prolong overall survival? How effective is it in controlling residual disease? What is the safety (side effects) of the treatment and how does it affect the patient's quality of life?

What participants need to do:

Be randomized to one of the treatment groups . Receive the appropriate treatment (maintenance therapy, or maintenance therapy plus radiotherapy) according to their group.

Have regular check-ups and imaging scans to assess the status of the tumor. Complete questionnaires about quality of life. May be asked to provide a blood sample for research . This study will help doctors to better understand how to treat this special group of patients with advanced lung cancer, with a view to improving their outcome and quality of life.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntary signed written informed consent and compliance with protocol requirements;
2. Age ≥ 18 years;
3. Expected survival time ≥ 3 months;
4. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1;
5. Histologically or cytologically confirmed advanced non-small cell lung cancer;
6. After receiving 4-6 cycles of first-line platinum-based chemotherapy combined with immunotherapy, PET-CT evaluation shows no disease progression, with no more than 5 lesions not meeting criteria for complete metabolic response, involving no more than 3 organs;
7. All residual lesions can safely receive radiation therapy as assessed by radiation oncologists;
8. Patient can tolerate the radiotherapy process, such as maintaining fixed position;
9. At least one measurable lesion among the oligoresidual lesions according to RECIST v1.1;
10. Agreement to provide archived tumor tissue specimens from primary or metastatic sites, or fresh tissue samples; if unable to provide tumor tissue samples, subjects may be enrolled after investigator assessment if meeting other inclusion/exclusion criteria;
11. Toxicities from previous anti-tumor therapies recovered to ≤ grade 1 per National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE v5.0) (excluding alopecia, fatigue, pigmentation, hypothyroidism stable on hormone replacement therapy, grade 2 peripheral neuropathy after chemotherapy, and exceptions specified in other inclusion criteria);
12. Laboratory values at screening must meet the following criteria: a) Neutrophils ≥ 1.5×10^9/L b) Platelets ≥ 100×10^9/L c) Hemoglobin ≥ 90g/L (no blood transfusion within 14 days) d) Serum Cr ≤ 1×ULN, endogenous creatinine clearance > 50ml/min (Cockcroft-Gault formula) e) AST ≤ 2.5×ULN; ALT ≤ 2.5×ULN; if liver metastases present, ALT and AST ≤ 5×ULN f) Total bilirubin ≤ 1.5×ULN (except for Gilbert's syndrome subjects, where total bilirubin must be < 51.3μmol/L) g) Thyroid Stimulating Hormone (TSH), Free Triiodothyronine (FT3), Free Thyroxine (FT4) all within ±10% of normal range.

Exclusion Criteria:

1. Archived tumor tissue, pre-treatment tumor biopsy, or histological examination showing evidence of previous small cell or mixed small cell/non-small cell histology;
2. Previous tissue samples or peripheral blood genetic sequencing reports indicating EGFR sensitizing mutations, ALK fusion, or other gene variations that should receive standard first-line targeted therapy; squamous cell carcinoma without genetic testing is presumed negative;
3. Symptomatic brain metastases;
4. Leptomeningeal metastases;
5. Active, known, or suspected autoimmune disease (excluding vitiligo, type I diabetes, residual hypothyroidism due to autoimmune thyroiditis requiring only hormone replacement therapy, or conditions not expected to recur in the absence of external triggers);
6. Active tuberculosis (TB) infection as determined by chest X-ray, sputum examination, and clinical examination. Patients with a history of active pulmonary TB infection within the previous year, even if treated, will be excluded. Patients with a history of active pulmonary TB infection more than 1 year ago will also be excluded unless effective previous anti-TB treatment can be documented;
7. Comorbidities requiring immunosuppressive medication, or requiring systemic or local use of corticosteroids at immunosuppressive doses;
8. Pregnancy or breastfeeding;
9. Interstitial lung disease with symptomatic manifestations, or that may interfere with the detection or management of suspected drug-related pulmonary toxicity;
10. Positive for human immunodeficiency virus antibody (HIVAb), active hepatitis B virus infection (HBsAg positive and HBV-DNA > 10^3 copies/ml), or hepatitis C virus infection (HCV antibody positive and HCV-RNA > lower limit of detection at the research center);
11. History of severe neurological or psychiatric disorders, including but not limited to: dementia, depression, seizures, bipolar disorder, etc.;
12. Receipt of other investigational drugs or treatments within 4 weeks prior to study randomization;
13. Use of any Chinese herbal medicines with anti-tumor activity within 2 weeks prior to study drug administration;
14. History of other malignancies (excluding non-melanoma skin cancer and the following in situ cancers: bladder, gastric, colon, endometrial, cervical/dysplasia, melanoma, or breast), unless complete remission was achieved at least 2 years prior to study enrollment and no additional therapy is required or anticipated during the study period;
15. History of severe cardiac or cerebrovascular disease, e.g., New York Heart Association (NYHA) ≥ class 2 heart failure, acute coronary syndrome (such as myocardial infarction, unstable angina, etc.) within 6 months of screening, acute cerebrovascular disease (such as transient ischemic attack, cerebral infarction, cerebral hemorrhage, etc.) within 6 months of screening;
16. Thromboembolic events requiring therapeutic intervention within 6 months prior to screening, such as unstable deep vein thrombosis, arterial thrombosis, and pulmonary embolism; excluding infusion-related thrombosis;
17. Planned vaccination or vaccination with live vaccines within 28 days prior to study randomization;
18. Other conditions deemed unsuitable for participation in this clinical trial by the investigator due to comorbidities or other circumstances.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 224 (Estimated)
Dates: Start 2025-06-11 (Actual); Primary Completion 2027-09-01 (Estimated); Study Completion 2027-09-01 (Estimated)

PRIMARY OUTCOMES:
Progression-Free Survival (PFS) | The estimated median PFS time from entry into maintenance therapy to recurrence in the control group is 6 months. The experimental group is expected to extend median PFS time from 6 months to 8.7 months.
  Time from randomization (with or without radiotherapy) to first occurrence of objective disease progression (Response Evaluation Criteria in Solid Tumors [RECIST] 1.1) or death from any cause (if occurring before disease progression).

CONTACTS AND LOCATIONS:
Overall Officials: Zhijie Wang, Study Director — Cancer Institute and Hospital, Chinese Academy of Medical Sciences
Locations (1):
- National Cancer Center/National Clinical Research Center for Cancer/Cancer Hospital, Chinese Academy of Medical Sciences and Peking Union Medical College, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sung H, Ferlay J, Siegel RL, Laversanne M, Soerjomataram I, Jemal A, Bray F. Global Cancer Statistics 2020: GLOBOCAN Estimates of Incidence and Mortality Worldwide for 36 Cancers in 185 Countries. CA Cancer J Clin. 2021 May;71(3):209-249. doi: 10.3322/caac.21660. Epub 2021 Feb 4. PMID 33538338
- [Background] Gao S, Li N, Wang S, Zhang F, Wei W, Li N, Bi N, Wang Z, He J. Lung Cancer in People's Republic of China. J Thorac Oncol. 2020 Oct;15(10):1567-1576. doi: 10.1016/j.jtho.2020.04.028. No abstract available. PMID 32981600
- [Background] Cheng Y, Zhang T, Xu Q. Therapeutic advances in non-small cell lung cancer: Focus on clinical development of targeted therapy and immunotherapy. MedComm (2020). 2021 Dec 14;2(4):692-729. doi: 10.1002/mco2.105. eCollection 2021 Dec. PMID 34977873
- [Background] Zappa C, Mousa SA. Non-small cell lung cancer: current treatment and future advances. Transl Lung Cancer Res. 2016 Jun;5(3):288-300. doi: 10.21037/tlcr.2016.06.07. PMID 27413711
- [Background] Parikh RB, Cronin AM, Kozono DE, Oxnard GR, Mak RH, Jackman DM, Lo PC, Baldini EH, Johnson BE, Chen AB. Definitive primary therapy in patients presenting with oligometastatic non-small cell lung cancer. Int J Radiat Oncol Biol Phys. 2014 Jul 15;89(4):880-7. doi: 10.1016/j.ijrobp.2014.04.007. Epub 2014 May 24. PMID 24867533
- [Background] Winegarden JD, Mauer AM, Otterson GA, Rudin CM, Villalona-Calero MA, Lanzotti VJ, Szeto L, Kasza K, Hoffman PC, Vokes EE; University of Chicago Phase II Network; Ohio State University. A phase II study of oxaliplatin and paclitaxel in patients with advanced non-small-cell lung cancer. Ann Oncol. 2004 Jun;15(6):915-20. doi: 10.1093/annonc/mdh215. PMID 15151948
- [Background] Guckenberger M, Lievens Y, Bouma AB, Collette L, Dekker A, deSouza NM, Dingemans AC, Fournier B, Hurkmans C, Lecouvet FE, Meattini I, Mendez Romero A, Ricardi U, Russell NS, Schanne DH, Scorsetti M, Tombal B, Verellen D, Verfaillie C, Ost P. Characterisation and classification of oligometastatic disease: a European Society for Radiotherapy and Oncology and European Organisation for Research and Treatment of Cancer consensus recommendation. Lancet Oncol. 2020 Jan;21(1):e18-e28. doi: 10.1016/S1470-2045(19)30718-1. PMID 31908301
- [Background] Hellman S, Weichselbaum RR. Oligometastases. J Clin Oncol. 1995 Jan;13(1):8-10. doi: 10.1200/JCO.1995.13.1.8. No abstract available. PMID 7799047
- [Background] Rim CH, Cho WK, Park S, Yoon WS, Yang DS. Role of local ablative treatment in oligometastatic non-small cell lung cancer: a meta-analysis. Int J Surg. 2023 Apr 1;109(4):1006-1014. doi: 10.1097/JS9.0000000000000339. PMID 36974686
- [Background] Dingemans AC, Hendriks LEL, Berghmans T, Levy A, Hasan B, Faivre-Finn C, Giaj-Levra M, Giaj-Levra N, Girard N, Greillier L, Lantuejoul S, Edwards J, O'Brien M, Reck M, Smit EF, Van Schil P, Postmus PE, Ramella S, Lievens Y, Gaga M, Peled N, Scagliotti GV, Senan S, Paz-Ares L, Guckenberger M, McDonald F, Ekman S, Cufer T, Gietema H, Infante M, Dziadziuszko R, Peters S, Porta RR, Vansteenkiste J, Dooms C, de Ruysscher D, Besse B, Novello S. Definition of Synchronous Oligometastatic Non-Small Cell Lung Cancer-A Consensus Report. J Thorac Oncol. 2019 Dec;14(12):2109-2119. doi: 10.1016/j.jtho.2019.07.025. Epub 2019 Aug 6. PMID 31398540
- [Background] Pawlik TM, Scoggins CR, Zorzi D, Abdalla EK, Andres A, Eng C, Curley SA, Loyer EM, Muratore A, Mentha G, Capussotti L, Vauthey JN. Effect of surgical margin status on survival and site of recurrence after hepatic resection for colorectal metastases. Ann Surg. 2005 May;241(5):715-22, discussion 722-4. doi: 10.1097/01.sla.0000160703.75808.7d. PMID 15849507
- [Background] Pastorino U, Buyse M, Friedel G, Ginsberg RJ, Girard P, Goldstraw P, Johnston M, McCormack P, Pass H, Putnam JB Jr; International Registry of Lung Metastases. Long-term results of lung metastasectomy: prognostic analyses based on 5206 cases. J Thorac Cardiovasc Surg. 1997 Jan;113(1):37-49. doi: 10.1016/s0022-5223(97)70397-0. PMID 9011700
- [Background] Franceschini D, De Rose F, Cozzi S, Franzese C, Rossi S, Finocchiaro G, Toschi L, Santoro A, Scorsetti M. The use of radiation therapy for oligoprogressive/oligopersistent oncogene-driven non small cell lung cancer: State of the art. Crit Rev Oncol Hematol. 2020 Apr;148:102894. doi: 10.1016/j.critrevonc.2020.102894. Epub 2020 Feb 5. PMID 32062314
- [Background] Kordbacheh T, Honeychurch J, Blackhall F, Faivre-Finn C, Illidge T. Radiotherapy and anti-PD-1/PD-L1 combinations in lung cancer: building better translational research platforms. Ann Oncol. 2018 Feb 1;29(2):301-310. doi: 10.1093/annonc/mdx790. PMID 29309540
- [Background] Pitroda SP, Chmura SJ, Weichselbaum RR. Integration of radiotherapy and immunotherapy for treatment of oligometastases. Lancet Oncol. 2019 Aug;20(8):e434-e442. doi: 10.1016/S1470-2045(19)30157-3. Epub 2019 Jul 29. PMID 31364595
- [Background] Van Limbergen EJ, De Ruysscher DK, Olivo Pimentel V, Marcus D, Berbee M, Hoeben A, Rekers N, Theys J, Yaromina A, Dubois LJ, Lambin P. Combining radiotherapy with immunotherapy: the past, the present and the future. Br J Radiol. 2017 Aug;90(1076):20170157. doi: 10.1259/bjr.20170157. Epub 2017 May 25. PMID 28541096
- [Background] Zhou Y, Yu F, Zhao Y, Zeng Y, Yang X, Chu L, Chu X, Li Y, Zou L, Guo T, Zhu Z, Ni J. A narrative review of evolving roles of radiotherapy in advanced non-small cell lung cancer: from palliative care to active player. Transl Lung Cancer Res. 2020 Dec;9(6):2479-2493. doi: 10.21037/tlcr-20-1145. PMID 33489808
- [Background] Ng CS, Wan IY, Yim AP. Impact of video-assisted thoracoscopic major lung resection on immune function. Asian Cardiovasc Thorac Ann. 2009 Aug;17(4):426-32. doi: 10.1177/0218492309338100. PMID 19713346